CLINICAL TRIAL: NCT02851940
Title: Pain and Bleeding Following Hypertonic Saline Sclerotherapy Compared to Brand Ligation for Symptomatic Hemorrhoids: A Randomized Prospective Study
Brief Title: Pain and Bleeding Following Hypertonic Saline Sclerotherapy Compared to Brand Ligation for Symptomatic Hemorrhoids
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients recruited
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM.FD.04
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2016-05

CONDITIONS: Hemorrhoids; Bleeding; Pain
Keywords: Pain; Bleeding; Hemorrhoids; Band Ligation; hypertonic saline sclerotherapy
MeSH Terms: conditions — Hemorrhoids; Hemorrhage; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Rubber Band Ligation) (Experimental): 15 patients
  Interventions: Procedure: Rubber Band Ligation
- B (Hypertonic Saline Infusion) (Experimental): 15 patients
  Interventions: Procedure: Hypertonic Saline Infusion

INTERVENTIONS:
Procedure: Rubber Band Ligation — Anoscopic rubber band ligation by bedside with patient in the jack-knife position (equipment: anoscope, rubber band applicator)
  Arms: A (Rubber Band Ligation)
Procedure: Hypertonic Saline Infusion — Endoscopic retroflexed 3 ml injection of 20% hypertonic saline 1cm above the dentate line (equipment: Flex sig, injection needle, 20% saline)
  Arms: B (Hypertonic Saline Infusion)

SUMMARY:
The investigators aim at prospectively comparing procedural pain, adverse events and rebleeding rates of anoscopic rubber band ligation and endoscopic hypertonic saline injection in patients with symptomatic hemorrhoidal disease

DETAILED DESCRIPTION:
Hemorrhoidal disease is a common encounter in a gastroenterologist's practice. These are often symptomatic, either bleeding or prolapsing. There are no set guidelines in our institution (The American University of Beirut Medical Center - AUBMC) for the treatment of symptomatic hemorrhoidal disease. Two types of treatment are available at our institution: anoscopic rubber band ligation (RBL) or endoscopic sclerotherapy (ESC) with hypertonic (20%) saline. Both methods have been shown to be effective in the literature, with above 75% complete symptomatic relief from a single application after 8-12 months. Post procedural pain of RBL in two randomized studies ranged 40-47%, while different studies showed post procedural pain following ESC to be 12-39%. However no study has ever compared these two therapeutic methods head-on, neither has any study compared both procedures for tolerability and rebleeding rates.

Research design and methods:

This study is a randomized, prospective study conducted at the American University of Beirut Medical Center which will involve 30 patients suffering from symptomatic hemorrhoidal disease requiring therapeutic intervention. Patients meeting inclusion criteria will be randomized using a computer generated randomization list to either Rubber Band Ligation (RBL) or Hypertonic Saline Sclerotherapy as a therapeutic interventional procedure.

- Patients will be approached by their Gastroenterologist during clinic visits and informed about the study. If participants wish to take part in the study, they will be given additional study information, screened for inclusion criteria, and consented by the research assistant or clinic nurse. Recruitment and randomization will occur during the same visit after patient consent in order to properly schedule patients for their therapeutic interventional procedures. All rubber band ligations will be performed by one endoscopist and all sclerotherapies will be performed by the other endoscopist.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Consent to the study
* Bleeding grade 1,2 and 3 hemorrhoids

Exclusion Criteria:

* Age under 18 years
* Refusal to sign consent
* Prior surgical and non surgical hemorrhoid procedure/manipulation
* External hemorrhoids
* Thrombosed hemorrhoids
* Active Anal Fissure
* Active anal fistula
* Immunocompromised
* Grade 4 internal hemorrhoids
* Chronic Pain requiring analgesics
* Antiplatelets and anticoagulation intake other than Aspirin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Composite Pain Score | Days 0 after procedure
  Range 0 (no pain) to 10 (maximum pain)
Composite Pain Score | Day 3 after procedure
  Range 0 (no pain) to 10 (maximum pain)
Composite Pain Score | Day 7 after procedure
  Range 0 (no pain) to 10 (maximum pain)

SECONDARY OUTCOMES:
Bleeding | Days 1 to 7 after the procedure
  If any bleeding is noticed upon defecation
Pain Medication Usage | Days 1 to 7 after the procedure
Bleeding | week 1-week 7 post procedure, 3 months, 6 months
  If any bleeding is noticed upon defecation
Pain | week 1-week 7 post procedure, 3 months, 6 months
  Range 0 (no pain) to 10 (maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Ala I Sharara, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
In the publication